CLINICAL TRIAL: NCT02955030
Title: Phase 1 Study to Determine the Safety and Immunogenicity of a Sublingual Administration of NSV0001 in Healthy Male Volunteers
Brief Title: Evaluation of the Safety and Immunogenicity of a Sublingual Influenza Vaccine NSV0001 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nitto Denko Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NSV0001-01
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- NSV0001(Cohort1) (Experimental): 15 µg of hemagglutinin [HA] antigen per strain with 150 µg of ND002 adjuvant, administration by sublingual route
  Interventions: Biological: NSV0001
- NSV0001(Cohort2) (Experimental): 30 µg of hemagglutinin[HA] antigen per strain with 300 µg of ND002 adjuvant, administration by sublingual route
  Interventions: Biological: NSV0001
- NSV0001(Cohort3) (Experimental): 60 µg of hemagglutinin[HA] antigen per strain with 600 µg of ND002 adjuvant, administration by sublingual route
  Interventions: Biological: NSV0001
- Placebo (Placebo Comparator): 0 µg of hemagglutinin[HA] antigen per strain with 0 µg of ND002 adjuvant, administration by sublingual route
  Interventions: Biological: Placebo
- Influenza HA vaccine "Biken HA" (Active Comparator): Seasonal quadrivalent influenza vaccine, administration by subcutaneous injection route
  Interventions: Biological: Influenza HA vaccine "Biken HA"

INTERVENTIONS:
Biological: NSV0001 — sublingual
  Arms: NSV0001(Cohort1); NSV0001(Cohort2); NSV0001(Cohort3)
Biological: Influenza HA vaccine "Biken HA" — subcutaneous
  Arms: Influenza HA vaccine "Biken HA"
Biological: Placebo — sublingual
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a sublingual administration of NSV0001 in healthy male volunteers.

DETAILED DESCRIPTION:
NSV0001 is a quadrivalent influenza vaccine with the new adjuvant (ND002) administered by sublingual route.

This study will enroll healthy male adults. Participants will receive two doses of the vaccine, 4 weeks apart, and will stay in the investigational site for 2 consecutive days after each vaccination.

Participants will keep a patient diary to record the local and systemic reactions for one week after each vaccination. In addition, the safety monitoring will be extended through 6 months from the last vaccination to detect the potential immune mediated disorders (pIMD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 20 to 49 years of age on the date of informed consent
2. Individuals who are determined eligible healthy adult to participate clinical study from the results of medical history, medical examination and clinical estimation by principal investigator / sub-investigator.
3. Written informed consent was obtained from the subject. And the subject whom principal investigator/ sub-investigator judged about the following conditions; the subject will be able to follow study instructions, subject will be able to receive medical examination and tests prescribed in the protocol and subject will be able to inform indication, etc.
4. Individuals who will be able to receive telephone communication during clinical trial participations

Exclusion Criteria:

1. History of administration of seasonal influenza HA vaccine within 180 days
2. History of infection of influenza within 180 days
3. History of receiving live attenuated vaccine within 28 days or inactivated vaccine/ toxoid within 7 days
4. History of receiving any of following treatment such as medical drugs I. Within 28 days: 1. Interferon products, 2. Drugs affected to immune system (e.g., immunosuppressant), 3. Systemic or inhalant adrenocorticosteroid, 4. G-CSF and M-CSF II. Within 84 days: 1. HGG products, 2. Blood products, 3. blood transfusion (including blood component transfusion) III. Within 180 days: 1. massive dose therapy of HGG products (≥200 mg/kg)
5. History of previous causing of anaphylaxis by intake of foods or drugs (including vaccine)
6. History of previous finding to be suspected allergic reaction of oral cavity, pharynx or laryngeal mucosa
7. Individuals who have hypersensitivity against seasonal influenza HA vaccine or chicken egg, chicken meat and other chicken derived materials
8. Individuals who have experience of fever more than 39.0℃ or finding to be suspected allergic reaction e.g. generalized rash within two days after previous preventive treatment (seasonal influenza vaccine and other vaccines)
9. History of anamnestic convulsion (excluding anamnestic fever convulsion in childhood)
10. History of previously diagnosis of immunodeficiency, or individuals who have close relatives (within third degree) with congenital immunodeficiency syndrome
11. History of anamnestic Guillain-Barre syndrome or ADE (Acute Disseminated Encephalomyelitis)
12. Individuals who have poorly controlled cardiovascular, hematological, hepatic, renal, gastrointestinal, urological or endocrine metabolic diseases, and such diseases possibly affect to the participation of clinical study or study results
13. Individuals who have respiratory diseases e.g. interstitial pneumonia and bronchial asthma
14. Individuals who is associated with allergic rhinitis, and have a symptom
15. Individuals who have experienced whole blood donation of not less than 400 mL within 12 weeks, whole blood donation of not less than 200 mL within 4 weeks, or apheresis within 2 weeks
16. Individuals who have received other study medication within 4 months
17. Individuals who have inflammation, swelling or uncomfortable feeling, or mechanical problem in oral cavity, sublingual, tongue, pharynx or laryngeal mucosa, which disturbing sublingual administration or affecting absorption
18. Individuals who have not recovered from injury of laryngeal mucosa caused by treatment of dental extraction etc. (excluding treatment of carious teeth)
19. Individuals who is associated with disease with abnormal salivation (Sjogren's syndrome, well-defined dry mouth / xerostomia etc.)
20. Individuals who have positive reaction against any of STS (serological test for syphilis) (TP antibody, lipid antibodies), HBs antigen, HCV antibody, or HIV antigen/ antibody
21. History of anamnestic drug abuse (defined as illegal drug use) or alcoholism within one year before IMP dosing, or individuals who will not give up consuming excessive alcohol
22. Individuals who have clinically problematic abnormality in 12-lead electrocardiogram in the examination
23. Individuals who have been found abnormal value in clinical laboratory tests, which suggesting clinically problematic complications, or individuals who have been found abnormal value in the following test items: ALT and/ or AST that is more than 3 times of the upper limit of standard value.
24. In addition, individuals whom principal investigator/ sub-investigator judged inappropriate as the subject of such clinical trial

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with local and systemic reactions and subjects reporting one or more adverse events | 28 days after last vaccination

SECONDARY OUTCOMES:
Seroconversion rate of serum HI antibody titer for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
GMT ratio of serum HI antibody titer for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
Reciprocal cumulative frequency distribution of serum HI antibody titer for each four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
Sero-protection rate of serum HI antibody titer for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
Seroconversion rate of serum neutralizing antibody titer for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
GMT ratio of serum neutralizing antibody for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination
Reciprocal cumulative frequency distribution of serum neutralizing antibody titer for each of four strains(A/H1N1, A/H3N2, B/Yamagata, and B/Victoria) | 28 days after last vaccination

OTHER OUTCOMES:
Change of immunological response of IgA ELISA specific for A/H1N1 in serum | 28 days after last vaccination
Change of immunological response of IgA ELISA specific for A/H1N1 in the nasal wash | 28 days after last vaccination
GMT ratio of immunological response of IgA ELISA specific for A/H1N1 in the nasal wash | 28 days after last vaccination
Change of immunological response of IgA ELISA specific for A/H1N1 in saliva | 28 days after last vaccination
GMT ratio of immunological response of IgA ELISA specific for A/H1N1 in saliva | 28 days after last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Senior fellow, Study Chair — Nitto Denko Corporation
Locations (1):
- OPHAC Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No